CLINICAL TRIAL: NCT01063595
Title: A Comparative, Open-label, Randomized, Cross-over Phase I Trial in Healthy Volunteers to Investigate the Relative Efficacy, Safety and Tolerability of Octaplas LG™ vs. Octaplas®
Brief Title: A Trial to Investigate the Relative Efficacy, Safety, and Tolerability of Octaplas LG Versus Octaplas SD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LAS-203
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Comparison of Octaplas LG and Octaplas SD
Keywords: Octaplas LG; Octaplas SD

ARMS (2):
- Octaplas LG (Experimental): Participants received 1200 mL of Octaplas LG intravenously once.
  Interventions: Biological: Octaplas LG
- Octaplas SD (Active Comparator): Participants received 1200 mL of Octaplas SD intravenously once.
  Interventions: Biological: Octaplas SD

INTERVENTIONS:
Biological: Octaplas LG — Octaplas LG was composed of human coagulation-active plasma treated with solvent/detergent for 1-1.5 hours to remove enveloped viruses, eg, HIV, HBV, and HCV. An additional manufacturing step, involving an affinity ligand gel, removed prion proteins. Octaplas LG was provided frozen in pyrogen free plastic bags.
  Arms: Octaplas LG
Biological: Octaplas SD — Octaplas SD was composed of human coagulation-active plasma treated with solvent/detergent for 4-4.5 hours to remove enveloped viruses, eg, HIV, HBV, and HCV. Octaplas SD was provided frozen in pyrogen free plastic bags.
  Arms: Octaplas SD

SUMMARY:
The primary objective of the study was to compare the efficacy of Octaplas LG with Octaplas SD in terms of recovery of coagulation factors and other haemostatic parameters. The secondary objective of the study was to compare the safety and tolerability of Octaplas LG with Octaplas SD in terms of haematological and clinical chemistry parameters and adverse event monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with all aspects of the protocol.
* Signed Informed Consent.
* Capable of understanding the plasmapheresis information sheet and sign it.
* Healthy male or female volunteers, age 18 years or older.
* Women must have negative pregnancy test (human chorionic gonadotropin [HCG] based assay).
* Women must have sufficient methods of contraception (eg, intrauterine device, oral contraception, etc).
* No clinically relevant abnormalities in medical history and general physical examination.
* Standard health insurance.

Exclusion Criteria:

* Pregnancy or lactation.
* Tattoos within the last 3 months.
* Subject was treated therapeutically with fresh frozen plasma, blood, or plasma-derived products within the last 6 months.
* Hypersensitivity to blood products or plasma proteins.
* History of angioedema.
* History of coagulation or bleeding disorder or any other known abnormality affecting coagulation, fibrinolysis, or platelet function.
* Any clinically significant abnormal laboratory values.
* IgA deficiency.
* Seropositivity for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus type 1 or type 2 antibodies.
* Symptoms of a clinically relevant illness within 3 weeks before the first trial day.
* History of or suspected drug or alcohol abuse.
* Subjects currently participating in another clinical study.
* Any investigational medicinal product administration within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology - Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Jilma-Stohlawetz P, Kursten FW, Horvath M, Leitner G, List J, Marcek J, Quehenberger P, Schwameis M, Bartko J, Derhaschnig U, Jilma B. Recovery, safety, and tolerability of a solvent/detergent-treated and prion-safeguarded transfusion plasma in a randomized, crossover, clinical trial in healthy volunteers. Transfusion. 2013 Sep;53(9):1906-17. doi: 10.1111/trf.12075. Epub 2013 Jan 16. PMID 23320451

RESULTS

PARTICIPANT FLOW:
Groups:
- Octaplas SD First, Then Octaplas LG: Participants received 1200 mL of Octaplas SD intravenously once. At least 4 weeks later, participants received 1200 mL of Octaplas LG intravenously once.
- Octaplas LG First, Then Octaplas SD: Participants received 1200 mL of Octaplas LG intravenously once. At least 4 weeks later, participants received 1200 mL of Octaplas SD intravenously once.
Period: Enrolled in Study and Randomized
Arm/Group | Octaplas SD First, Then Octaplas LG | Octaplas LG First, Then Octaplas SD
Started | 32 | 31
Received Treatment | 31 | 29
Completed | 31 | 29
Not Completed | 1 | 2
Not completed — Reason not Specified | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawn by the Investigator | 0 | 1
Period: First Intervention
Arm/Group | Octaplas SD First, Then Octaplas LG | Octaplas LG First, Then Octaplas SD
Started | 31 | 29
Completed | 29 | 24
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Reason not Specified | 0 | 1
Period: Second Intervention
Arm/Group | Octaplas SD First, Then Octaplas LG | Octaplas LG First, Then Octaplas SD
Started | 29 | 24
Completed | 29 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least 1 of the study treatments in any study period.
Groups:
- All Participants: Participants received 1200 mL of Octaplas LG intravenously once and 1200 mL of Octaplas SD intravenously once in a crossover design.
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Recovery of the Coagulation Factors I, II, V, VII, VIII, IX, X, and XI
Description: Recovery was defined as the maximum percentage change of the coagulation factor value measured 5 minutes after the end of plasmapheresis to the coagulation factor value measured at 15 minutes or 2 hours after the end of study drug administration. The coagulation parameters were measured by validated assays from blood samples obtained 5 minutes after the end of plasmapheresis and 15 minutes and 2 hours after the end of study drug administration.
Time Frame: From 5 minutes after the end of plasmapheresis up to 2 hours after the end of study drug administration
Population: Per protocol population: All participants who had evaluable efficacy measurements in both of the treatment periods.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Octaplas LG | Octaplas SD
Number analyzed (Participants) | 43 | 43
Percentage change
  Factor I | 8.11 (8.93) | 9.12 (8.75)
  Factor II | 7.08 (6.46) | 6.68 (7.35)
  Factor V | 6.31 (9.35) | 6.91 (10.09)
  Factor VII | 8.48 (11.03) | 9.28 (14.53)
  Factor VIII | 1.50 (9.38) | 5.21 (9.93)
  Factor IX | 8.86 (9.11) | 11.08 (7.74)
  Factor X | 7.90 (8.96) | 9.97 (12.37)
  Factor XI | 6.53 (6.32) | 8.24 (7.54)

2. Primary Outcome: Recovery of the Haemostatic Parameters Prothrombin Time, Activated Partial Thromboplastin Time, and Protein C
Description: Recovery was defined as the maximum (minimum for activated partial thromboplastin time) percentage change of the haemostatic parameter value measured 5 minutes after the end of plasmapheresis to the haemostatic parameter value measured at 15 minutes or 2 hours after the end of study drug administration. The haemostatic parameters were measured by validated assays from blood samples obtained 5 minutes after the end of plasmapheresis and 15 minutes and 2 hours after the end of study drug administration.
Time Frame: From 5 minutes after the end of plasmapheresis up to 2 hours after the end of study drug administration
Population: Per protocol population: All participants who had evaluable efficacy measurements in both of the treatment periods.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Octaplas LG | Octaplas SD
Number analyzed (Participants) | 43 | 43
Percentage change
  Prothrombin time | 1.36 (4.71) | 2.85 (6.18)
  Activated partial thromboplastin time | -4.60 (3.71) | -5.73 (4.39)
  Protein C | 9.49 (8.44) | 9.75 (6.97)

3. Secondary Outcome: Concentration of Plasmin Inhibitor
Description: Values of plasmin inhibitor were measured by validated assays from blood samples obtained 30 minutes before plasmapheresis, 5 minutes after the end of plasmapheresis, 15 minutes and 2 hours after the end of study drug administration, and 24 hours and 7 days after initiation of plasmapheresis. The concentration of plasmin inhibitor is reported as the percentage of plasmin inhibition. A higher concentration of plasmin inhibitor results in a higher percentage of plasmin inhibition.
Time Frame: From 30 minutes before plasmapheresis up to 24 hours after the end of plasmapheresis
Population: Per protocol population: All participants who had evaluable efficacy measurements in both of the treatment periods.
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Octaplas LG | Octaplas SD
Number analyzed (Participants) | 43 | 43
Percentage inhibition
  Pre-plasmapheresis 30 minutes | 90.51 (9.93) | 91.53 (9.12)
  Post-plasmapheresis 5 minutes | 85.72 (9.34) | 85.67 (10.08)
  Post-transfusion 15 minutes | 79.81 (8.15) | 74.93 (8.72)
  Post-transfusion 2 hours | 79.21 (8.45) | 75.23 (9.11)
  Post-plasmapheresis 24 hours | 88.35 (9.41) | 85.40 (8.93)
  Post-plasmapheresis 7 days | 90.95 (9.79) | 91.65 (9.88)

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 of the study treatments in any study period.
Arm/Group | Octaplas LG | Octaplas SD
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 34/60 | 39/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octaplas LG (N=60) | Octaplas SD (N=60)
Anaphylactic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octaplas LG (N=60) | Octaplas SD (N=60)
Nausea (Gastrointestinal disorders) | 3 | 1
Urticaria (Immune system disorders) | 10 | 9
Headache (Nervous system disorders) | 8 | 9
Paraesthesia (Nervous system disorders) | 3 | 2
Paraesthesia oral (Nervous system disorders) | 9 | 6
Vertigo (Nervous system disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No